CLINICAL TRIAL: NCT03881072
Title: Evaluating the Endometrial Receptivity of FET Patients by Ultrasounicelastography and Predicting the Pregnancy Outcome.
Brief Title: Evaluating the Endometrial Receptivity of FET Patient by Ultrasounicelastography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Bing Yao, Professor，Chief physician, Jinling Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UE evaluating Em-receptivity
Record Dates: First submitted 2018-09-12; First posted 2019-03-19 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Assisted Reproductive Technology; Ultrasonography
Keywords: Ultrasounicelastography; Frozen embryo transplantation; Endometrial Receptivity; pregnancy outcome

STUDY DESIGN:
Intervention Model Description: Prospective study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultrasounicelastography (Other): Ultrasounicelastography:non-invasive, convenient and comprehensive evaluation method.
  Interventions: Other: Ultrasounicelastography

INTERVENTIONS:
Other: Ultrasounicelastography — Observing the correlation between endometrial elasticity score, endometrial blood flow index (PI, RI, S/D, endometrial thickness, morphology) and clinical pregnancy rate.

SUMMARY:
Prospective clinical study ：observing the correlation between endometrial elasticity score, endometrial blood flow index (PI, RI, S/D, endometrial thickness, morphology) and clinical pregnancy rate. In order to find a non-invasive, convenient and comprehensive evaluation method of evaluating the endometrial receptivity, and to provide effective means for the frozen embryo transplantation patients to improving pregnancy outcome.

DETAILED DESCRIPTION:
Randomly selecting 20-40 years patients were prepared to accept frozen embryo transplant ; HRT cycle preparation of endometrium；choosing HRT plan to prepare the transplantation endometrium.Establishing a strict standard of exclusion and exclude standard to exclude endometrial lesions and underlying disease.The patients were given elastography for 5-7 days afterEndometrium transformation.Observing the correlation between endometrial elasticity score, endometrial blood flow index (PI, RI, S/D, endometrial thickness, morphology) and clinical pregnancy rate. In order to find a non-invasive, convenient and comprehensive evaluation method of evaluating the endometrial receptivity, and to provide effective means for the frozen embryo transplantation patients to improving pregnancy outcome.

ELIGIBILITY:
Inclusion Criteria:

1. the volunteers voluntarily signed the informed consent.
2. female patients between 20-40 years old.
3. HRT cycle.
4. no uterine cavity operation was performed within 3 months.

Exclusion Criteria:

1. endometrial polyps, abnormal uterine cavity, intrauterine adhesions and dysplasia of uterus.
2. hydrosalpinx was not ligated.
3. patients with uterine myoma and uterine fibroids;

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-01-10 (Actual); Study Completion 2018-12-10 (Actual)

PRIMARY OUTCOMES:
endometrial receptivity | Month 12
  Observing the correlation between elasticity score, endometrial blood flow index (PI, RI, S/D, endometrial thickness, morphology) and clinical pregnancy rate.

CONTACTS AND LOCATIONS:
Locations (1):
- Yao Bing, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
In order to find a non-invasive, convenient and comprehensive evaluation method of evaluating the endometrial receptivity, and to provide effective means for the frozen embryo transplantation patients to improving pregnancy outcome.